CLINICAL TRIAL: NCT02946658
Title: Use of Autologous, Adult Adipose-Derived Stem/Stromal Cells (AD-cSVF) in Chronic Lung Disorders
Brief Title: Use of Autologous, Adult Adipose-Derived Stem/Stromal Cells In Chronic Lung Disorders
Acronym: ADcSVF-COPD
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID-19 stopped patient ability to complete access for outcome analysis
Sponsor: Healeon Medical Inc (Industry)
Collaborators: Terry, Glenn C., M.D. (Individual)
Responsible Party: Principal Investigator, Robert W. Alexander, MD, FICS, Principal Investigator, Science, Healeon Medical Inc
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGV-GARM 2
Record Dates: First submitted 2016-10-03; First posted 2016-10-27 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Lung Disease
Keywords: COPD, Emphysema
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lipoaspiration Arm 1 (Experimental): Acquisition of Adipose-Derived tissue Stromal Vascular Fraction (AD-tSVF) via closed syringe harvest subdermal fat
  Interventions: Procedure: lipoaspiration
- AD-cSVF Arm 2 (Experimental): Isolation of cellular stem/stromal cells from subdermal adipose-derived cellular stromal vascular fraction (AD-cSVF)
  Interventions: Procedure: ADcSVF
- Normal Saline IV Arm 3 (Experimental): Normal Saline IV with AD-cSVF cells
  Interventions: Procedure: Normal Saline IV

INTERVENTIONS:
Procedure: lipoaspiration — Closed syringe harvesting subdermal fat
  Arms: Lipoaspiration Arm 1
Procedure: ADcSVF — Isolation of AD-cSVF
  Arms: AD-cSVF Arm 2
Procedure: Normal Saline IV — Normal Saline IV containing AD-cSVF
  Arms: Normal Saline IV Arm 3

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a lung-related disorder that is characterized by long-term, often progressive state of poor airflow. Primary symptoms include low oxygen tension, shortness of breath, productive cough, and broncho-pulmonary inflammation and interference with oxygen-carbon dioxide exchange.

Air pollution and tobacco smoking are felt to be the most common cause of these issues. Diagnostic testing is based on poor airflow measured by lung function studies and whose symptoms do not improve much with antiasthma bronchodilators.

Study is an interventional study to document the safety and efficacy of use of AD-cSVF in chronic broncho-pulmonary disease groups.

DETAILED DESCRIPTION:
COPD is often treated by limiting exposure to poor air quality, but there is no cure at this time. Attempted therapy include smoking cessation, vaccinations, respiratory rehabilitation, and attempts of use of bronchodilators and steroids. Many resort to supplemental oxygen therapy, lung transplantation, and antibiotic supportive therapy during exacerbations.

As of 2013, COPD involve approximately 5% pf the global populations (approximately 330 million). Most commonly it occurs approximately equally between men/women and result in about 3 million deaths per year. Estimates of economic costs are estimated to be more than 2.1 trillion dollars in 2010.

This study includes microcannula harvesting of subdermal adipose tissues, incubation, digestion and isolation of AD-cSVF. This stromal cellular pellet (without actual extracellular matrix or stromal elements) is then suspended in 500 cc sterile Normal Saline (NS) and deployed via peripheral intravenous route. Evaluations of safety issues are measured at intervals (both severe and non-severe categories) and by repeated pulmonary function studies.

ELIGIBILITY:
Inclusion Criteria:

* Prior Diagnosis of moderate to severe COPD
* GOLD II a, III, IV

Exclusion Criteria:

* Pregnant or Lactating Females
* Life expectancy of < 3 months due to concomitant illnesses
* Exposure to any investigational drug or procedure with 1 month prior to study entry or enrollment in concurrent study which may interfere with interpretation of study results
* Illness which, in investigators judgement, may interfere with the patient' ability to comply with protocol, compromise patient safety, ability to provide informed consent to study, or interfere with interpretation of study outcomes
* Subjects on chronic immunosuppressive or chemotherapeutic medications
* Known drug or alcohol dependence or other factors which may interfere with study conduct or interpretation of result or in the opinion of investigator are not suitable to participate.
* Subjects with documented Alpha-1 Antitrypsin Deficiency (Inherited lung and liver disorder)
* Unwilling or not competent to understand and execute an informed consent agreement
* Patients positive for Hepatitis (Hepatitis A history excepted)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2026-08-14 (Estimated); Study Completion 2027-08-14 (Estimated)

PRIMARY OUTCOMES:
Safety - Pulmonary Function | 12 months Evaluate Function and Adverse Events
  Pulmonary Function to be Addressed as occurrence or frequency of adverse event during study

SECONDARY OUTCOMES:
Change from Baseline Respiratory Rate | 1 month, 6 month, 1 year
  Measured rate clinically at rest
GOLD Classification | 1 year
  Global Initiative for Chronic Obstructive Lung Disease (GOLD) is a COPD staging system based on degree of airflow limitations (obstruction) and measured by pulmonary function studies
Change from baseline 6 Minute Walk Test | 12 Months
  Exercise capacity measured by distance a patient can walk in 6 minute timeframe
Change from Baseline Lung X-Ray | 6 months, 12 months
  standard flat film x-ray
Change from Baseline SGOT Blood Testing | 1 Month
  Measure Blood Serum Glutamate Oxaloacetate Transaminase (SGOT) Measure Blood Elevation with liver damage
Change from Baseline SGPT Blood Testing | 1 Month
  Measure Blood Serum Glutamate Pyruvate Transaminase (SGPT) elevation with liver damage
Pulmonary Function Testing | Baseline, 6 Months
  Measure Baseline Pulmonary Function (FEV/FEVi Measure)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Alexander, MD, Principal Investigator — Healeon Medical Inc; Glenn C. Terry, MD, Principal Investigator — Global Alliance for Regenerative Medicine (GARM)
Locations (2):
- Regenevita LLC, Stevensville, Montana, United States
- Global Alliance for Regenerative Medicine (GARM), Roatán, HN, Honduras

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Decramer M, Janssens W, Miravitlles M. Chronic obstructive pulmonary disease. Lancet. 2012 Apr 7;379(9823):1341-51. doi: 10.1016/S0140-6736(11)60968-9. Epub 2012 Feb 6. PMID 22314182
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Mahler DA. Mechanisms and measurement of dyspnea in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2006 May;3(3):234-8. doi: 10.1513/pats.200509-103SF. PMID 16636091
- [Background] Holland AE, Hill CJ, Jones AY, McDonald CF. Breathing exercises for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD008250. doi: 10.1002/14651858.CD008250.pub2. PMID 23076942
- [Background] Kennedy SM, Chambers R, Du W, Dimich-Ward H. Environmental and occupational exposures: do they affect chronic obstructive pulmonary disease differently in women and men? Proc Am Thorac Soc. 2007 Dec;4(8):692-4. doi: 10.1513/pats.200707-094SD. PMID 18073405
- [Background] Devereux G. ABC of chronic obstructive pulmonary disease. Definition, epidemiology, and risk factors. BMJ. 2006 May 13;332(7550):1142-4. doi: 10.1136/bmj.332.7550.1142. No abstract available. PMID 16690673
- [Background] Foreman MG, Campos M, Celedon JC. Genes and chronic obstructive pulmonary disease. Med Clin North Am. 2012 Jul;96(4):699-711. doi: 10.1016/j.mcna.2012.02.006. Epub 2012 Mar 6. PMID 22793939
- [Background] Brode SK, Ling SC, Chapman KR. Alpha-1 antitrypsin deficiency: a commonly overlooked cause of lung disease. CMAJ. 2012 Sep 4;184(12):1365-71. doi: 10.1503/cmaj.111749. Epub 2012 Jul 3. No abstract available. PMID 22761482
- [Background] O'Donnell DE. Hyperinflation, dyspnea, and exercise intolerance in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2006 Apr;3(2):180-4. doi: 10.1513/pats.200508-093DO. PMID 16565429
- [Background] Mackay AJ, Hurst JR. COPD exacerbations: causes, prevention, and treatment. Med Clin North Am. 2012 Jul;96(4):789-809. doi: 10.1016/j.mcna.2012.02.008. Epub 2012 Mar 16. PMID 22793945
- [Background] Puhan MA, Gimeno-Santos E, Scharplatz M, Troosters T, Walters EH, Steurer J. Pulmonary rehabilitation following exacerbations of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD005305. doi: 10.1002/14651858.CD005305.pub3. PMID 21975749
- [Background] Saxena A, Watkin SW. Bilateral malignant testicular carcinoid. Br J Urol. 1990 Mar;65(3):302-3. doi: 10.1111/j.1464-410x.1990.tb14738.x. No abstract available. PMID 2337756
- [Background] Kew KM, Seniukovich A. Inhaled steroids and risk of pneumonia for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2014 Mar 10;2014(3):CD010115. doi: 10.1002/14651858.CD010115.pub2. PMID 24615270
- [Background] COPD Working Group. Long-term oxygen therapy for patients with chronic obstructive pulmonary disease (COPD): an evidence-based analysis. Ont Health Technol Assess Ser. 2012;12(7):1-64. Epub 2012 Mar 1. PMID 23074435
- [Background] Bradley JM, O'Neill B. Short-term ambulatory oxygen for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD004356. doi: 10.1002/14651858.CD004356.pub3. PMID 16235359
- [Background] Vollenweider DJ, Jarrett H, Steurer-Stey CA, Garcia-Aymerich J, Puhan MA. Antibiotics for exacerbations of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Dec 12;12:CD010257. doi: 10.1002/14651858.CD010257. PMID 23235687
- [Background] Inamdar AC, Inamdar AA. Mesenchymal stem cell therapy in lung disorders: pathogenesis of lung diseases and mechanism of action of mesenchymal stem cell. Exp Lung Res. 2013 Oct;39(8):315-27. doi: 10.3109/01902148.2013.816803. Epub 2013 Aug 30. PMID 23992090
- [Background] Conese M, Piro D, Carbone A, Castellani S, Di Gioia S. Hematopoietic and mesenchymal stem cells for the treatment of chronic respiratory diseases: role of plasticity and heterogeneity. ScientificWorldJournal. 2014 Jan 19;2014:859817. doi: 10.1155/2014/859817. eCollection 2014. PMID 24563632
- [Background] McQualter JL, Anthony D, Bozinovski S, Prele CM, Laurent GJ. Harnessing the potential of lung stem cells for regenerative medicine. Int J Biochem Cell Biol. 2014 Nov;56:82-91. doi: 10.1016/j.biocel.2014.10.012. Epub 2014 Oct 15. PMID 25450456
- [Background] Tzouvelekis A, Ntolios P, Bouros D. Stem cell treatment for chronic lung diseases. Respiration. 2013;85(3):179-92. doi: 10.1159/000346525. Epub 2013 Jan 29. PMID 23364286
- [Background] Tzouvelekis A, Laurent G, Bouros D. Stem cell therapy in chronic obstructive pulmonary disease. Seeking the Prometheus effect. Curr Drug Targets. 2013 Feb;14(2):246-52. doi: 10.2174/1389450111314020009. PMID 23256721